CLINICAL TRIAL: NCT04224545
Title: Colchicine for Prevention Atrial Fibrillation After Cardiac Surgery in the Early Postoperative Period
Brief Title: COlchicine in Cardiac Surgery
Acronym: COCS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bakulev Scientific Center of Cardiovascular Surgery (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #2.20122019
Record Dates: First submitted 2019-12-27; First posted 2020-01-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Colchicine Adverse Reaction; Atrial Fibrillation New Onset
Keywords: Colchicine; Postoperative atrial fibrillation; Anti-inflammatory; Cardiac surgery; Sympatholytic
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: A randomized double-blind controlled trial in two groups
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental): Colchicine 1 mg day (COLCHICINA LIRCA ® ACARPIA Farmaceutici S.r.l.)
  Interventions: Drug: Colchicine Pill
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine Pill — Colchicine at a dose of 1 mg a day before surgery, 2, 3, 4, 5 days after surgery.
  Other Names: group C
  Arms: Colchicine
Drug: Placebo — Placebo started a day before surgery, 2, 3, 4, 5 days after surgery.
  Other Names: group P
  Arms: Placebo

SUMMARY:
Postoperative atrial fibrillation (POAF) is a major complication of cardiac surgery, which could lead to high morbidity and mortality, increase duration of hospital stay and increase the cost of treatment. Colchicine possesses both anti-inflammatory and sympatholytic properties, so it has been studied to prevent POAF. The ACC/AHA guidelines for colchicine contain a class IIB recommendation, but the ESC guidelines do not recommend this drug. More researches are needed to focus on reducing of side effects by optimizing the colchicine regimen to reduce the incidence of gastrointestinal side effects. It is believed that further research is needed to investigate the efficacy and safety of colchicine in these conditions.

This research is aimed to study the effectiveness of short-term administration of the drug.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF) is a major complication of cardiac surgery, which could lead to high morbidity and mortality, increase duration of hospital stay and increase the cost of treatment. Postoperative AF is considered as a multifactorial phenomenon. Its pathogenesis is characterized by inflammation, oxidative stress and autonomic dysfunction. Several predisposing factors lead to the development of POAF, including pre -, intra-and postoperative factors. The main of them are age, previous history of major cardiovascular risk factors and ischemic reperfusion injury during surgery. Treatment of POAF involves drugs to control the frequency of rhythm in hemodynamically stable patients and other treatment regimens usually used for the treatment of AF. Intraoperative administration of beta-blockers and some antiarrhythmic drugs is recommended by international clinical guidelines. In addition, previous treatment consisting of the use of colchicine, magnesium sulfate, statins and antioxidants have reduced the incidence of postoperative AF. However, the results of large-scale randomized trials have observed the development of undesirable adverse reactions.

Despite these recommendations, the question of the correct regimen for prevention of POAF remains controversial. Colchicine possesses both anti-inflammatory and sympatholytic properties, so it has been studied to prevent POAF. The ACC/AHA guidelines for colchicine contain a class IIB recommendation, but the ESC guidelines do not recommend this drug.

Two studies sequentially COPPS-1 and COPPS-2 evaluated the effect of colchicine on the incidence of POAF after open heart surgery (COPPS-1) and the development of postcardiotomy syndrome (COPPS-2). In COPPS-1, patients (n=336) were treated with colchicine from the third day after surgery for a month and showed a significant decrease of POAF after heart surgery over the entire follow-up period. 360 patients were evaluated in the COPPS-2 study. The incidence of POAF between the colchicine and placebo groups was comparable, although colchicine significantly reduced postpericardiotomy syndrome. The main limitation of the COPSS-2 study was the high rate of cessation of intervention (20% of participants), which had a significant impact on the outcome of the trial.

Based on the latest meta-analysis of the colchicine effect on POAF after heart surgery, it was found that it still reduces POAF compared with control (HR = 0.69, 95% IM 0.57-0.84, p = 0.0002) and the duration of hospital stay was reduced by 1.2 days (95% IM -1.89 to -0.44, p = 0.002); however, the frequency of adverse gastrointestinal events increased significantly (HR = 2.52, 95% IM 1.62-3.93, p < 0.0001). Despite the high level of side effects, a significant reduction of POAF outweighs the balance in the favor of its use. However, more researches are needed to focus on reducing of side effects by optimizing the colchicine regimen to reduce the incidence of gastrointestinal side effects. It is believed that further research is needed to investigate the efficacy and safety of colchicine in these conditions.

This research is aimed to study the effectiveness of short-term administration of the drug.

ELIGIBILITY:
Inclusion Criteria:

Adult patients awaiting elective cardiac surgery (CABG and/or AVR (aortic valve replacement), who are willing and able to give informed consent for participation in the study and who are in sinus rhythm and not taking any antiarrhythmic medication, except beta-adrenergic blocking agents, at the time before surgery.

Exclusion Criteria:

* History of persistent or long-term atrial fibrillation/atrial flutter
* Congenital heart disease, except the bicuspid AV
* Frequent VE/SVE, AV block 2-3 degrees
* Use of corticosteroids during the last month
* Taking any antiarrhythmic drugs, except beta-blockers, within the last 1 month
* Prior "open" heart surgery
* Moderate to severe renal failure (creatinine clearance < 50 ml / min)
* History of obstructive hepato-biliary disease or other serious hepatic disease
* Significant mitral valve disease (moderate or severe mitral regurgitation-eg. > grade II and/or mitral stenosis & mitral annular calcification).
* Patient participation in another clinical trial

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative atrial fibrillation. | Monitoring is carried out immediately after surgery and will be continued until the end of the 7th postoperative day.
  POAF detected on continuous ECG monitoring.

SECONDARY OUTCOMES:
Number of participants with lethal and non-lethal events. | Participants will be followed for the duration of the postoperative period up to the day of initial discharge from the hospital, an expected average of 7 days.
  The main nosocomial lethal and non-lethal events (death, stroke, myocardial infarction, heart failure).
Fluid in the pericardium. | Diagnostics will be carried out on the 3rd and 5th day after surgery.
  Fluid in the pericardium evaluated by echocardiography.
Fluid in the pleura. | Diagnostics will be carried out on the 3rd and 5th day after surgery.
  Fluid in the pleura evaluated by echocardiography.
Acute kidney damage (according to the dynamics of creatinine clearance). | Diagnostics will be carried out a day before surgery and on the 3rd and 5th day after surgery.
  Dynamics of creatinine clearance.
Inflammation in blood plasma. | Diagnostics will be carried out a day before surgery and on the 3rd and 5th day after surgery.
  Dynamics of biomarker of inflammation in blood plasma (neutrophils).
Liver damage | Diagnostics will be carried out a day before surgery and on the 3rd and 5th day after surgery.
  Dynamics of biomarkers of liver damage (aspartate aminotransferase, alanine aminotransferase).

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Shvartz, Principal Investigator — Bakulev National Medical Research Center for Cardiovascular Surgery
Locations (2):
- Russia (2):
  - Federal Center for Cardiovascular Surgery (Astrakhan), Astrakhan
  - Bakulev National Medical Research Center for Cardiovascular Surgery, Moscow

IPD SHARING:
Plan to Share IPD: Yes
The datasets analyzed during the current study are publicly available. The data is available in the general repository "Open Science Framework" at the link
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: until 2045
Access Criteria: open access
URL: https://doi.org/10.17605/OSF.IO/HPCZW

REFERENCES:
- [Result] Shvartz V, Le T, Kryukov Y, Sokolskaya M, Ispiryan A, Khugaeva E, Yurkulieva G, Shvartz E, Petrosyan A, Bockeria L, Bockeria O. Colchicine for Prevention of Atrial Fibrillation after Cardiac Surgery in the Early Postoperative Period. J Clin Med. 2022 Mar 3;11(5):1387. doi: 10.3390/jcm11051387. PMID 35268478
- [Result] Shvartz V, Le T, Enginoev S, Sokolskaya M, Ispiryan A, Shvartz E, Nudel D, Araslanova N, Petrosyan A, Donakanyan S, Chernov I, Bockeria L, Golukhova E. Colchicine in Cardiac Surgery: The COCS Randomized Clinical Trial. J Cardiovasc Dev Dis. 2022 Oct 20;9(10):363. doi: 10.3390/jcdd9100363. PMID 36286314
- [Result] Shvartz V.A., Le T.G., Enginoev S.T., Sokolskaya M.A., Ispiryan A.Yu., Shvartz E.N., Nudel D.V., Araslanova N.Kh., Petrosyan A.D., Talibova S.M., Donakanyan S.A., Chernov I.I., Boсkeria L.A., Golukhova E.Z. Association of new markers of systemic inflammation with the risk of developing for the first time postoperative atrial fibrillation when using colchicine in patients undergoing open heart surgery. Annals of arrhythmology. 2023; 20(1): 22-33. (In Russian).
- Available data/document: Individual Participant Data Set — https://doi.org/10.17605/OSF.IO/HPCZW — The datasets analyzed during the current study are publicly available. The data is available in the general repository "Open Science Framework" at the link